CLINICAL TRIAL: NCT02244879
Title: Effects of Resveratrol on Inflammation in Type 2 Diabetic Patients. A Double-blind Randomized Controlled Trial
Brief Title: Effects of Resveratrol on Inflammation in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Simona Bo, Dr, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RF-2010-2313155
Record Dates: First submitted 2014-09-15; First posted 2014-09-19 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes Mellitus; Inflammation; Insulin Resistance; Other Disorders of Bone Density and Structure
Keywords: resveratrol; type 2 diabetes mellitus; inflammation; insulin resistance; body composition; bone mass
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation; Insulin Resistance | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo (Placebo Comparator): In this arm, 64 patients will receive a tablet of placebo once/day for 6 months
  Interventions: Dietary Supplement: resveratrol
- resveratrol 40 (Experimental): In this arm, 64 patients will receive a tablet of 40mg resveratrol once/day for 6 months
  Interventions: Dietary Supplement: resveratrol
- resveratrol 500 (Experimental): In this arm, 64 patients will receive a tablet of 500 mg resveratrol once/day for 6 months
  Interventions: Dietary Supplement: resveratrol

INTERVENTIONS:
Dietary Supplement: resveratrol — arm resveratrol 500: 6 months of resveratrol 500 mg/day arm resveratrol 40: 6 months of resveratrol 40 mg/day

SUMMARY:
This research will investigate the effect of resveratrol on inflammatory mediators in type 2 diabetic patients in vivo.

The investigators will also investigate the hypothesis that resveratrol has an antioxidant activity, improves insulin sensitivity and lipid pattern, down-regulates bone-turnover.

DETAILED DESCRIPTION:
Despite a large body of evidence demonstrating promising effects of resveratrol in rodents, human studies are still lacking and both preventive and therapeutic value of resveratrol in humans remains to be elucidated. The published evidence is not sufficiently strong to recommend for the administration of resveratrol to humans, beyond dietary sources. On the other hand, animal data are promising in prevention of various cancer types, coronary heart diseases and diabetes which strongly indicate the need for human clinical trials.

Furthermore, data are lacking either about safety during long-term administration, or on the efficacy of resveratrol administration in patients with chronic illnesses, such as diabetes mellitus.

The main objective of this study is to investigate the effect of resveratrol on inflammatory mediators in type 2 diabetic patients in vivo.

This research will investigate the hypothesis that resveratrol, when given orally to type 2 diabetic subjects for 24 weeks induces a decrease in values of high-sensitivity CRP (C-reactive protein) (primary outcome measure), IL-6 (Interleukin-6), PTX3 (pentraxin 3).

The investigators will also investigate the hypothesis that resveratrol has an antioxidant activity, improves insulin sensitivity and lipid pattern, down-regulates bone-turnover. Secondary outcomes are therefore variations in the following variables: TAS (total antioxidant status), glycemia, glycated hemoglobin (HbA1c), Homeostasis model assessment of insulin resistance (HOMA-IR), total and HDL-cholesterol, triglycerides, adiponectin, body composition (evaluated by Dual-emission X-ray absorptiometry DXA-), bone mineral density (DXA).

Finally, the investigators are interested in evaluating efficacy, safety and tolerability of two different dosages of resveratrol: 500 mg/day and 40 mg/day.

ELIGIBILITY:
Inclusion Criteria:

1. 35 years of age and older
2. Type 2 diabetes with body mass index (BMI)<35 kg/m2
3. Subjects on hypoglycemic agents other than insulin
4. Willing to give written informed consent and able to understand, to participate in and to comply with the study requirements.

Exclusion Criteria:

1. Subjects on any antioxidant medication
2. Patient on non-steroidal anti-inflammatory drug, steroids or insulin
3. On any agent with significant antioxidant properties
4. History of drug or alcohol abuse
5. Liver or kidney diseases
6. Any life threatening diseases
7. Allergy to peanuts, grapes, wine, mulberries
8. Pregnant women
9. Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass surgery or coronary angioplasty) in the previous four Weeks
10. Subjects on anticoagulants

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
C reactive protein (CRP) | up to 25 months
  To investigate changes from baseline in blood concentrations of high-sensitivity CRP after six months of treatment with either resveratrol at different dosages or placebo

SECONDARY OUTCOMES:
Metabolic and oxidative markers | up to 25 months
  To evaluate before-after changes in the concentrations of the following: Interleukin 6, Pentraxin-3, total antioxidant status, fasting glucose, insulin, glycated hemoglobin, total and HDL-cholesterol, triglycerides, adiponectin.

OTHER OUTCOMES:
body composition and bone mineral density | up to 25 months
  To evaluate before-after change in bone mineral density and body composition by Dual-emission X-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Simona Bo, MD, Principal Investigator — University of Turin, Italy
Locations (1):
- University of Turin, Turin, IT, Italy

REFERENCES:
- [Derived] Bo S, Togliatto G, Gambino R, Ponzo V, Lombardo G, Rosato R, Cassader M, Brizzi MF. Impact of sirtuin-1 expression on H3K56 acetylation and oxidative stress: a double-blind randomized controlled trial with resveratrol supplementation. Acta Diabetol. 2018 Apr;55(4):331-340. doi: 10.1007/s00592-017-1097-4. Epub 2018 Jan 12. PMID 29330620
- [Derived] Bo S, Ponzo V, Evangelista A, Ciccone G, Goitre I, Saba F, Procopio M, Cassader M, Gambino R. Effects of 6 months of resveratrol versus placebo on pentraxin 3 in patients with type 2 diabetes mellitus: a double-blind randomized controlled trial. Acta Diabetol. 2017 May;54(5):499-507. doi: 10.1007/s00592-017-0977-y. Epub 2017 Feb 25. PMID 28238190